CLINICAL TRIAL: NCT00363961
Title: Resistance Training During Maintenance Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Carmen Castaneda Sceppa, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R03DK064825 (NIH); R03DK064825 (NIH)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; Maintenance dialysis; Resistance exercise; Muscle wasting; Disability
MeSH Terms: conditions — Kidney Failure, Chronic; Muscular Atrophy | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): resistance exercise
  Interventions: Behavioral: Resistance exercise
- 2 (Sham Comparator): flexibility exercises
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — resistance exercise vs sham comparison
  Other Names: strength training

SUMMARY:
There is a rising incidence of kidney failure in the US, with poor outcomes and high cost. End-stage renal disease (ESRD) affects almost 375,000 individuals in the US at a cost of more than $14 billion per year. Despite advances in dialysis and transplantation therapies, kidney failure leads to poor outcomes, poor prognosis and high health care costs. Malnutrition and the underlying systemic inflammatory response developed during the course of chronic kidney disease, worsen during ESRD, and lead to adverse outcomes, increased morbidity and mortality. Muscle wasting, impaired functional capacity and poor quality of life are the most important factors associated with malnutrition and inflammation in renal failure. We have shown in pre dialysis patients with moderate chronic renal insufficiency that the anabolic effects of resistance exercise training result in significant improvements in protein utilization, nutritional status and functional capacity even in the context of anorexia and prescribed low protein diets. Therefore, we propose to develop, test and implement a progressive resistance exercise routine for ESRD patients during the hemodialysis session. By implementing such intervention, we hope to offer a therapeutic strategy that can be incorporated to the standard of care of ESRD patients by working in conjunction with the dialysis unit staff.

DETAILED DESCRIPTION:
The hypotheses to be investigated are that, compared to ESRD patients on maintenance dialysis receiving stretches only, the addition of 30-45 min of progressive resistance training during the hemodialysis session will counteract the burden of renal disease and will result in:

1. A feasible and safe exercise modality for ESRD patients.
2. Will contribute to improved nutritional status and reduced systemic inflammation
3. Will result in improved quality of life

ELIGIBILITY:
Inclusion Criteria:

* Male and female ESRD patients over 30 years of age
* ESRD patients undergoing maintenance hemodialysis 3x/wk for at least 3 months
* Willing to be randomized to either study group
* Compliance with at least 80% of the dialysis sessions

Exclusion Criteria:

* Unstable cardiovascular disease
* Any uncontrolled chronic condition
* Cardiac surgery, myocardial infarction, joint replacement, or low extremity fracture within the previous 6 months
* Severe cognitive impairment resulting in inability to understand and provide written informed consent form and or follow instructions
* Current resistance training
* Low extremity amputees

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
- Physical function (short physical performance battery) | 6 months

SECONDARY OUTCOMES:
Muscle mass, inflammation biomarkers, quality of life(SF36), and Activities of Daily Living | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Castaneda-Sceppa, MD, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States